CLINICAL TRIAL: NCT06756321
Title: An Exploratory Clinical Study of the Safety and Efficacy of Chimeric Antigen Receptor T-Cells (CAR T-Cells) in Subjects with Relapsed/Refractory Hematologic Malignancy
Brief Title: A Study of CAR T-Cells in Relapsed/Refractory Hematologic Malignancy
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Affiliated Hospital of Nantong University (Other)
Collaborators: Shanghai First Song Biotechnology Co., LTD (Industry)
Responsible Party: Principal Investigator, Hong Liu, Chief of the Division of Hematology, Affiliated Hospital of Nantong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: X01-CN-A1
Record Dates: First submitted 2024-12-16; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Relapsed/refractory Lymphoma; Relapsed/Refractory Leukemia
MeSH Terms: conditions — Lymphoma; Leukemia | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cyclophosphamide + Fludarabine + CAR T-Cells (Experimental): Investigational product: anti-CD19-CAR T-cells, anti-CD30-CAR T-cell, anti-CD20/CD30-CAR T-cells.
  Subjects with CD19+ ALL or NHL will be infused with anti-CD19-CAR T-cells.
  Subjects with CD30+ HL or T-cell lymphoma will be infused with anti-CD30-CAR T-cells.
  Subjects with CD20+ lymphoma or CD20/CD30 double positive lymphoma who have relapsed after anti-CD19-CAR T-cell therapy will be infused with anti-CD20/CD30-CAR T-cells.
  Route of administration: Intravenous injection.
  Lymphodepleting chemotherapy regimen: A combination of fludarabine and cyclophosphamide will be administered prior to the infusion of CAR T-cells.
  Interventions: Biological: anti-CD19-CAR T-cells, or anti-CD30-CAR T-cells, or anti-CD20/CD30-CAR T-cells; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: anti-CD19-CAR T-cells, or anti-CD30-CAR T-cells, or anti-CD20/CD30-CAR T-cells — Each subject will be infused with single dose. A classic "3+3" dose escalation will be employed.
  anti-CD19-CAR T-cells
  Dose level 1：1x10^5 CAR T cells/kg, Dose level 2：3x10^5 CAR T cells/kg, Dose level 3：1x10^6 CAR T cells/kg
  anti-CD30-CAR T-cells
  Dose level 1：3x10^6 CAR T cells/kg, Dose level 2：6x10^6 CAR T cells/kg, Dose level 3：1x10^7 CAR T cells/kg
  anti-CD20/CD30-CAR T-cells
  Dose level 1：1x10^6 CAR T cells/kg, Dose level 2：3x10^6 CAR T cells/kg, Dose level 3：1x10^7 CAR T cells/kg
Drug: Fludarabine — Fludarabine will be given at a dose of 25 mg/m^2/day intravenously (IV) for 3 days prior to the infusion of CAR T-cells.
Drug: Cyclophosphamide — Cyclophosphamide will be given at a dose of 250 mg/m^2/day intravenously (IV) for 3 days prior to the infusion of CAR T-cells.

SUMMARY:
This study is a single-center, open-label clinical trial of single-dose of CAR T-cells in subjects with relapsed/refractory hematologic malignancy.

DETAILED DESCRIPTION:
The study will enroll subjects with relapsed/refractory hematologic malignancy, including lymphoma and leukemia. Subjects will receive a single infusion of CAR T-cells after screening, PBMC collection, and lymphodepleting chemotherapy. Toxicity will be assessed according to the Common Terminology Criteria for Adverse Events (CTCAE, version 5.0) from the National Cancer Institute. Safety of CAR T-cell therapy will be evaluated through laboratory tests, including 12-lead electrocardiograms, vital sign checks, and physical examination etc. Additionally, blood samples will be collected to study cellular pharmacokinetics and explore the effects of cell therapy on ferritin, C-reactive protein, and relevant cytokines.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following criteria to be eligible for the study:

  1. Voluntarily participate in the clinical study. The individual or the legal guardian fully understands the study, sign the informed consent form (ICF), and is willing and able to follow and complete all trial procedures.
  2. Age ≥ 18 years and < 70 years.
  3. Subjects with refractory or relapsed disease after current standard treatments (including allogeneic or autologous hematopoietic stem cell transplantation) who are not suitable for other treatment options, such as a second stem cell transplant. The definitions of relapsed/refractory lymphoma include one of the following situations:

     a. Relapsed/refractory B-cell acute lymphoblastic leukemia (ALL) is defined as one of the following:

     i) Primary refractory disease.

     ii) First relapse if the initial remission is ≤ 12 months.

     iii) Relapse or refractory disease after two or more lines of systemic therapy.

     iv) Relapse or refractory disease after allogeneic transplantation, provided that at the time of enrollment, the subject is at least 100 days post-stem cell transplantation and has not received immunosuppressive drugs for at least 4 weeks prior to enrollment, except for low-dose steroids (≤ 5 mg of prednisone or equivalent).

     b. Subjects with Ph+ B-cell ALL, who are intolerant to or ineligible for tyrosine kinase inhibitor (TKI) treatment, or who have relapsed/refractory disease after receiving at least two different TKI treatments, are eligible.

     c. Relapsed/refractory B-cell-derived non-Hodgkin lymphoma (NHL) and Hodgkin lymphoma (HL) defined as one of the following:

     i) No response to first-line treatment (primary refractory disease, excluding subjects intolerant to first-line treatment);
     * Disease progression (PD) as assessed after first-line treatment.
     * Best response of SD after at least 4 cycles of first-line treatment (e.g., 4 cycles of RCHOP), with SD duration not exceeding 6 months after the last dose.

     ii) No response to second-line or more treatments.
     * PD as the best response to the most recent treatment regimen.
     * Best efficacy of the last line of treatment as SD after at least 2 cycles, with the duration of SD not exceeding 6 months after the last dose.

     iii) Refractory after autologous stem cell transplant (ASCT).
     * Disease progression or relapse ≤ 12 months post-ASCT (relapsed patients must have biopsy-proven relapse).
     * If salvage treatment is performed after ASCT, the subjects must have no response to or relapsed after the last line of treatment.
     * Relapsed or refractory disease after two or more lines of systemic therapy.
  4. Indications included for enrollment in the cohort of anti-CD19-CAR T-cells:

     1. CD19+ ALL patients, with bone marrow smear reports showing tumor cells ≥ 5%.
     2. CD19+ NHL patients meeting one of the following subtypes:

        * Diffuse large B-cell Lymphoma, not otherwise specified (DLBCL-NOS)
        * Primary mediastinal B-cell lymphoma (PMBCL)
        * Transformed follicular lymphoma (TFL), previously treated for follicular lymphoma and then transformed to refractory DLBCL
        * Mantle cell lymphoma
        * High-grade B-cell lymphoma
        * Chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL)
  5. Subtypes of lymphoma included for enrollment in the cohort of anti-CD20/30-CAR T-cells:

     * Previously received anti-CD20/30-CAR T-cell therapy, with CD20 expression positive at enrollment.
     * Lymphoma with dual positive expression of CD20/CD30.
  6. Indications included for enrollment in the cohort of anti-CD30-CAR T-cell:

     * CD30 positive HL
     * CD30 positive T-cell lymphoma
  7. ECOG performance status ≤ 2.
  8. Expected survival of at least 12 weeks.
  9. Adequate venous access (for apheresis) and no other contraindications for blood cell separation.
  10. Laboratory tests during screening must meet the following requirements, and the subject must not have received cell growth factors (long-acting colony-stimulating factors (G-CSF/PEG-CSF) require a 2-week interval) and platelet transfusions within 7 days prior to hematological assessment:

      1. Absolute neutrophil count ≥ 1.0×10^9/L (the condition of ALL patients is determined by the investigator).
      2. Hemoglobin ≥ 60 g/L (without red blood cell transfusion in the last 14 days).
      3. Platelets ≥ 50×10^9/L (the condition of ALL patients is determined by the investigator).
      4. Absolute lymphocyte count (ALC) ≥ 0.5×10^9/L.
      5. Total serum bilirubin ≤ 1.5× the upper limit of normal (ULN).
      6. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5×ULN.
      7. Creatinine <1.5×ULN and estimated creatinine clearance ≥60 mL/min.
  11. Ejection fraction ≥ 45%, with echocardiogram (ECHO) confirming no pericardial effusion (excluding small or physiological amounts), and electrocardiogram results with no clinical significance.
  12. Baseline oxygen saturation > 92% without supplemental oxygen.
  13. Women of childbearing potential must have a negative serum or urine pregnancy test result (women who have undergone surgical sterilization or have been postmenopausal for at least 2 years are not considered of childbearing potential).

Exclusion Criteria:

* Subjects are not eligible to participate in this study if they meet any of the following criteria:

  1. ALL patients with central nervous system (CNS) abnormalities, including CNS-2 and CNS-3 that are of clinically significant neurological changes:

     1. CNS-3 disease is defined as detectable tumor cells in the cerebrospinal fluid (CSF) sample with ≥ 5 WBCs/mm^3, with or without neurological changes.
     2. CNS-2 disease is defined as detectable tumor cells in the CSF sample with < 5 WBCs/mm^3 and with neurological changes.

     Note: Subjects classified as CNS-1 (no detectable tumor cells in CSF) and those with no clinically significant neurological changes classified as CNS-2 are eligible to participate in this study.
  2. Brain MRI evidence shows central nervous system lymphoma. Active primary central nervous system DLBL, unless CNS involvement has been effectively treated (i.e., participants are asymptomatic) and there has been a local treatment interval of >4 weeks prior to enrollment.
  3. Presence of active central nervous system diseases, such as epilepsy, cerebrovascular ischemia/hemorrhage, dementia, cerebellar diseases, or any autoimmune diseases with CNS involvement.
  4. A history of or concurrent presence of other malignancies.
  5. Clinically significant cardiac disease or arrhythmias that cannot be controlled with medication.
  6. Presence or suspicion of fungal, bacterial, viral, or other infections that are uncontrolled or require intravenous antibiotics for treatment. Uncomplicated urinary tract infections and uncomplicated bacterial pharyngitis are allowed.
  7. Positive for hepatitis B (positive for HBsAg, and/or positive for Hepatitis B core antibody and HBV DNA >1000 copies/mL) and hepatitis C (positive for HCV antibodies), syphilis or human immunodeficiency virus (HIV) infection.
  8. Presence of any indwelling or drainage catheters (such as percutaneous nephrostomy tubes, indwelling Foley catheters, bile drainage tubes, or pleural/peritoneal/pericardial catheters). The use of specialized central venous access devices, such as Port-A-Cath® or Hickman® catheters, is allowed.
  9. Prior medication:

     1. Use of clofarabine or cladribine within 3 months prior to enrollment, or use of PEG-asparaginase within 3 weeks prior to enrollment.
     2. Injection of live vaccines within 4 weeks prior to enrollment.
     3. Donor lymphocyte infusion (DLI) within 28 days prior to enrollment.
     4. Any medications used for the treatment of GVHD (such as calcineurin inhibitors, methotrexate, mycophenolate, rapamycin, thalidomide) within 4 weeks prior to enrollment, or immunosuppressive antibodies (such as anti-CD20, anti-tumor necrosis factor, anti-interleukin-6, or anti-interleukin-6 receptor) used within 4 weeks prior to enrollment.
     5. Immune stimulation or immunosuppressive therapy (such as interferon-α, interferon-β, IL-2, etanercept, infliximab, tacrolimus, cyclosporine, or mycophenolic acid) within 4 weeks prior to enrollment.
     6. Any systemic immunosuppressive/stimulatory checkpoint molecule therapy within 4 weeks prior to enrollment (such as ipilimumab, nivolumab, pembrolizumab, atezolizumab, OX40 agonists, 4-1BB agonists, etc.).
     7. Use of systemic cytotoxic drugs within 2 weeks prior to enrollment, including daily or weekly low-dose maintenance chemotherapy (such as cyclophosphamide, ifosfamide, bendamustine, chlorambucil, methotrexate, vincristine, etc.).
     8. Long-acting growth factors (e.g., pegylated filgrastim) within 14 days prior to leukapheresis, or short-acting growth factors or mobilizing agents (e.g., granulocyte colony-stimulating factor/filgrastim, plerixafor) within 5 days prior to leukapheresis.
     9. Radiation therapy within 2 weeks prior to enrollment.
     10. Use of pharmacological doses of corticosteroids (>5 mg/day of prednisone or equivalent doses of other corticosteroids) and other immunosuppressive medications must be avoided within 7 days prior to enrollment.
     11. Use of venetoclax (BCL-2 inhibitor) within 4 days prior to leukapheresis.
     12. Short-acting targeted therapy (e.g., tyrosine kinase inhibitors) within 72 hours prior to leukapheresis.
     13. Idelalisib (oral PI3Kδ inhibitor) within 2 days prior to leukapheresis.
     14. Lenalidomide within 1 day prior to leukapheresis.
  10. Active graft-versus-host disease (GVHD) ≥ grade 2 on the CIBMTR acute GVHD grading system or requires systemic steroids at doses greater than physiological levels.
  11. A history of autoimmune diseases (such as Crohn's disease, rheumatoid arthritis, or systemic lupus) resulting in end-organ injury or requiring systemic immunosuppression/systemic disease-modifying agents within the last 2 years.
  12. A history of myocardial infarction, cardiac angioplasty or stenting, unstable angina, or other clinically significant cardiac diseases within 12 months prior to enrollment.
  13. A history of a concomitant genetic syndrome associated with bone marrow failure such as Fanconi anemia, Kostmann syndrome, and Shwachman-Diamond syndrome.
  14. A history of symptomatic deep vein thrombosis or pulmonary embolism requiring systemic anticoagulation within 6 months prior to enrollment. Subjects need to be on preventive anticoagulant medication.
  15. A history of other malignancies (except for non-melanoma skin cancer, in situ breast/cervical cancer, and other malignant tumors that have been effectively controlled without treatment in the past five years).
  16. Use of other investigational products within 30 days prior to screening.
  17. Pregnant or breastfeeding women of childbearing age. Chemotherapy poses potential risks to the fetus or infant. Women who have undergone surgical sterilization or are postmenopausal for at least 2 years are not considered of childbearing potential.
  18. Male and female subjects unwilling to practice birth control from the time of consent through 12 months after the completion of lymphodepleting chemotherapy or CAR T cells infusion (whichever is longer).
  19. Any medical activities that may interfere with the safety or efficacy assessment of the study treatment.
  20. In the investigator's judgment, the subject is unlikely to complete all protocol-required procedures and follow-up visits, or to comply with the requirements for participating in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2025-03-18 (Estimated); Study Completion 2026-03-18 (Estimated)

PRIMARY OUTCOMES:
Evaluate safety and tolerability of CAR T-cells | 28 days after infusion of CAR T-cells
  Proportion of subjects experiencing dose-limiting toxicities (DLT)
Evaluate the feasibility of administration of CAR T-cells | 12 months
  The proportion of subjects for whom the desired dose of CAR T-cells can be successfully manufactured

SECONDARY OUTCOMES:
Adverse events | 12 months
  Will be assessed using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0. AEs will be summarized in terms of type (organ affected or laboratory determination), severity, time of onset, duration, probable association with the study treatment and reversibility or outcome.
Incidence of cytokine release syndrome (CRS) and neurotoxicity | 12 months
  Will be assessed using ASTCT Criteria.
Evaluate cellular kinetics and persistence of CAR T-cells | 28 days after CAR T infusion, after which the evaluation is at the discretion of investigator
  Test Copy number of CAR in peripheral blood
Preliminary anti-tumor effect | 12 months
  Efficacy evaluation will be based on the National Comprehensive Cancer Network guidelines version 1. 2022 (ALL), or Lugano criteria (Lymphoma)
Overall response rate (ORR) | 12 months
  Overall response rate (ORR) defined as proportion of subjects achieving partial response or better
Progression-free survival (PFS) | Up to 1 year after CAR-T infusion
  Progression-free survival（PFS） defined as the time from the date of CAR T infusion to the first assessment of confirmed disease progression or death, whichever occurs first.
Overall survival (OS) | Up to 15 years after CAR-T infusion
  Overall survival defined as the time from the date of CAR T infusion of the subject to death due to any cause
Evaluate host immunogenicity to CAR T-cells | 12 months
  Incidence of anti-scFv antibodies
Evaluate toxicology of CAR T-cells | 28 days after CAR T infusion, after which the evaluation is at the discretion of investigator
  Levels of cytokines in serum, including IL-6, IL-10, IFN-γ, TNF-α

CONTACTS AND LOCATIONS:
Overall Officials: Hong Liu, MD, Principal Investigator — Affiliated Hospital of Nantong University
Locations (1):
- Affiliated Hospital of Nantong University, Nantong, Jiangsu, China

REFERENCES:
- [Derived] Huang Y, Gong Y, Liu X, Ruan H, Lu J, Kouros-Mehr H, Liu H, Wang H. Case Report: Bispecific CD20/CD30-targeted chimeric antigen receptor T-cell therapy for non-Hodgkin's lymphoma. Front Immunol. 2025 May 8;16:1567149. doi: 10.3389/fimmu.2025.1567149. eCollection 2025. PMID 40406106